CLINICAL TRIAL: NCT03485976
Title: Ixekizumab in the Treatment of Pityriasis Rubra Pilaris (PRP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Teri Greiling, Assistant Professor of Dermatology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018031
Record Dates: First submitted 2018-03-20; First posted 2018-04-03 (Actual); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Pityriasis Rubra Pilaris
Keywords: Ixekizumab; IL-17; Pityriasis Rubra Pilaris (PRP)
MeSH Terms: conditions — Pityriasis Rubra Pilaris | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ixekizumab treatment arm (Experimental): Ixekizumab 160 mg subcutaneous injection at week 0, followed by 80 mg subcutaneous injections at week 2, 4, 6, 8, 10, 12, 16, and 20
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Treatment at the FDA-approved psoriasis dosing
  Other Names: Taltz; IL-17A inhibitor

SUMMARY:
15 patients with PRP will be treated with ixekizumab for 24 weeks to determine safety and efficacy. Participants are required to travel to Portland, OR only for the first visit and week-24 visit. 5 visits in between these times and one follow up visit may be performed by secure videoconferencing.

DETAILED DESCRIPTION:
Pityriasis rubra pilaris (PRP) is a rare and poorly understood severe inflammatory skin disease characterized by widespread (often full-body) redness and flaking of the skin, painful thickening and cracking of the palms and soles, hair loss, crumbling nails, and severe skin itching and burning.

There is no FDA-approved therapy for this rare disease and the commonly used medications do not work for many patients. There is some evidence that IL-17 may be too high in the skin of PRP patients. Ixekizumab is an injectable medication that blocks IL-17 and is FDA-approved for psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PRP by clinical assessment and biopsy.
* Male subject age 18-99.
* Female subject age 18-99; either of non-childbearing potential or of childbearing potential who test negative for pregnancy and agree to use a reliable method of birth control or remain abstinent during the study and for at least 12 weeks following the last dose of ixekizumab.
* PASI score of 10 or greater at baseline.
* Are a candidate for phototherapy and/or systemic therapy.
* Willingness to travel to OHSU for all study visits, OR living >30 miles from OHSU and willing/able to participate in remote videoconferencing visits with access to a computer with internet capabilities and webcam.
* Have given written informed consent approved by the OHSU Investigational Review Board.

Exclusion Criteria:

* Known malignancy or lymphoproliferative disease (except treated basal cell skin cancer, treated squamous cell skin cancer, or treated cervical carcinoma in situ) for at least 5 years.
* Active, untreated, acute or chronic infection (such as untreated tuberculosis), or immunocompromised to an extent that such that participation in the study would pose an unacceptable risk to the subject. (Treated infections such as latent tuberculosis after completion of the appropriate therapy are not excluded.)
* Positive for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
* Previous treatment with any agent that targets interleukins 17 specifically.
* Systemic treatment or phototherapy for PRP within the past 4 weeks or 5 half-lives prior to baseline, whichever is longer. For biologic therapies, the specific washout periods used will be: etanercept <28 days; infliximab, adalimumab, or alefacept <60 days; golimumab <90 days; ustekinumab <8 months; rituximab or efalizumab <12 months.
* Have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the subject if participating in this study.
* Have a live vaccine within 12 weeks prior to baseline or intend to have a live vaccine during the course of study.
* Had any major surgery within 8 weeks prior to baseline or will require major surgery during the study that, in the opinion of the investigator, would pose an unacceptable risk to the subject.
* Presence of significant uncontrolled cerebrovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or neuropsychiatric disorders, or abnormal laboratory screening values that, in the opinion of the investigator, pose an unacceptable risk to the subject if participating in the study or of interfering with the interpretation of the data.
* Presence of inflammatory bowel disease
* Have clinical laboratory test results at screening that are outside the normal reference range of the population and are considered clinically significant, or have any of the following specific abnormalities: Neutrophil count <1500 cells/µL, lymphocyte count <500 cells/µL, platelet count <100,000 cells/µL, AST or ALT > 2.5 times the upper limit of normal, hemoglobin <8.5 g/dL for male subjects and <8.0 g/dL for female subjects, serum creatinine >2.0 mg/dL.
* Women who are lactating or breastfeeding.
* Have any other condition that precludes the subject from following and completing the protocol, in the opinion of the investigator.
* Are investigator site personnel directly affiliated with this study and/or their immediate families (spouse, parent, child, or sibling).

Are currently enrolled in, or discontinued from a clinical trial involving an investigational product or non-approved use of a drug or device within the last 4 weeks or a period of at least 5 half-lives of the last administration of the drug, whichever is longer, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teri Greiling, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haynes D, Strunck JL, Topham CA, Ortega-Loayza AG, Kent G, Cassidy PB, Hu R, Choate K, Wang Z, Liu Y, Greiling TM. Evaluation of Ixekizumab Treatment for Patients With Pityriasis Rubra Pilaris: A Single-Arm Trial. JAMA Dermatol. 2020 Jun 1;156(6):668-675. doi: 10.1001/jamadermatol.2020.0932. PMID 32293641

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixekizumab Treatment Arm
Started | 12
Completed | 11
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients at baseline
Arm/Group | Ixekizumab Treatment Arm
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 44.8 [23.2 to 73.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 28.0 [19.4 to 44.6]
PRP Subtype [Count of Participants; unit: Participants] — PRP can be categorized into six different subtypes based on age, duration, and pattern of skin involvement. Subtypes I and II generally occur in adulthood with a generalized skin rash; subtypes III, IV, and V are seen in children and adolescents; subtype VI is associated with HIV infection.
  The subtypes can be categorized as follows: Classic Adult (Type I); Atypical Adult (Type II); Classic Juvenile (Type III); Circumscribed Juvenile (Type IV); Atypical Juvenile (Type V); HIV-associated (Type VI)
  Participants
    Classic adult (Type I PRP) | 6
    Atypical adult (Type II PRP) | 5
    Classic juvenile (Type III PRP) | 1
Psoriasis Assessment and Severity Index (PASI) score [Median (Full Range); unit: units on a scale] — The psoriasis assessment and severity index (PASI) is a scale that measures the severity of skin disease by evaluating the redness, scale, and elevation of each body surface area of skin involved in psoriasis (a disease that has some similarities with PRP). Redness, scale, and elevation are each scored on a 0-4 point scale, added together, and multiplied by each body surface area involved (head and neck, trunk, upper limbs, lower limbs). The maximum score is 72 which would indicate the worst disease over every surface of someone's body. A scale of zero would indicate normal skin.
  units on a scale | 24.8 [12.6 to 57.6]
Physician Global Assessment (PGA) score [Count of Participants; unit: Participants] — The Physician Global Assessment (PGA) score is clinician-assessed 5-point scoring system used to assess overall disease severity. Scores range from 0 to 4, with higher numbers reflecting more severe disease. The scoring system is as follows:
  Clear (0); Almost clear (1); Mild (2); Moderate (3); Severe (4)
  Participants
    Clear (0) | 0
    Almost clear (1) | 0
    Mild (2) | 0
    Moderate (3) | 9
    Severe (4) | 3
Dermatology Life Quality Index (DLQI) score [Median (Full Range); unit: units on a scale] — The Dermatology Life Quality Index (DLQI) is a patient-administered survey that assesses impacts of disease on quality of life. There are 10 questions covering symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question refers to the impact of PRP on the patient's life over the previous week. The highest score is 30 and would indicate a maximum (negative) impact on quality of life. A score of zero would indicate no impact on quality of life.
  units on a scale | 19 [9 to 28]
Itch Numerical Rating Score (NRS) [Median (Full Range); unit: units on a scale] — The itch numerical rating score (NRS) is a patient reported measure of itch which is assessed on a 10-point scale. The scores range from a minimum score of 0 (no itch) to a maximum score of 10 (worst itch imaginable), with higher numbers reflecting more severe itch.
  units on a scale | 7 [4 to 10]
Pain Numerical Rating Score (NRS) [Median (Full Range); unit: units on a scale] — The pain numerical rating score (NRS) is a patient reported measure of pain which is assessed on a 10-point scale. The scores range from a minimum score of 0 (no pain) to a maximum score of 10 (worst pain imaginable), with higher numbers reflecting more severe pain.
  units on a scale | 6 [3 to 9]
Age at PRP diagnosis [Median (Full Range); unit: years] | 43.7 [10.3 to 73.0]
Duration of PRP symptoms prior to trial enrollment [Median (Full Range); unit: months] | 11.9 [1.4 to 453.8]
Previous systemic therapy [Number; unit: participants]
  Treatment naive | 1
  Prior systemic therapy | 11
  Prior methotrexate | 6
  Prior systemic retinoid | 7
  Prior biologic therapy | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement in PRP Severity and Body Surface Area
Description: Clinical improvement will be measured by the Psoriasis Area and Severity Index (PASI) score. PASI is a scale that measures the severity (redness, scale, and elevation) of each body surface area of skin involved in psoriasis (a disease that has some similarities with PRP). Redness, scale, and elevation are each scored on a 0-4 point scale, added together, and multiplied by each body surface area involved (head and neck, trunk, upper limbs, lower limbs). The maximum score is 72 which would indicate the worst disease over every surface of someone's body. A scale of zero would indicate normal skin.
Time Frame: 24 weeks
Population: Mean improvement in PASI from baseline to week-24
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab Treatment Arm
Number analyzed (Participants) | 12
units on a scale | 15.2 (2.1)
Statistical Analysis 1: Comparison: Ixekizumab Treatment Arm; Test type: Other; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05

2. Secondary Outcome: Improvement in Quality of Life
Description: Quality of life will be measured by the Dermatology Life Quality Index (DLQI). There are 10 questions covering symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question refers to the impact of PRP on the patient's life over the previous week. The highest score is 30 and would indicate a maximum (negative) impact on quality of life. A score of zero would indicate no impact on quality of life.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab Treatment Arm
Number analyzed (Participants) | 12
units on a scale | 9.5 (2.5)
Statistical Analysis 1: Comparison: Ixekizumab Treatment Arm; Test type: Other; p = 0.004, t-test, 2 sided — The threshold for significance was p=0.05

3. Secondary Outcome: Improvement in Itch
Description: Itch will be measured using a numeric rating scale from 0 (no itch) to 10 (worst itch imaginable).
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Ixekizumab Treatment Arm
Number analyzed (Participants) | 12
units on a scale | 3.6 (0.8)
Statistical Analysis 1: Comparison: Ixekizumab Treatment Arm; Test type: Other; p = 0.001, t-test, 2 sided — Threshold for significance was p=0.05

ADVERSE EVENTS:
Time Frame: 24-weeks
Arm/Group | Ixekizumab Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab Treatment Arm (N=12)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Gastrointestinal upset (Gastrointestinal disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Temporary worsening of PRP (Skin and subcutaneous tissue disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Ingrown nail (Skin and subcutaneous tissue disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Non-specific chest pain (resolved without intervention) (Cardiac disorders) | 1 (1)
Mild leukopenia (Blood and lymphatic system disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Cutaneous atrophy associated with corticosteroid use (Skin and subcutaneous tissue disorders) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03485976/Prot_SAP_000.pdf